CLINICAL TRIAL: NCT03100435
Title: Efficacy of Er:YAG Laser in Decontamination of Dental Implants: An In-Vitro Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Robert Gyurko, DMD, PhD, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12380
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: All participants will wear a mouth guard holding 8 titanium discs for 3 days, during which time a natural bacterial biofilm will form on the disc surfaces. After 3 days, the discs will be removed from the mouthguard, and treated ex vivo with different decontamination methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Er:YAG Laser (Experimental): Er:YAG Laser only
  Interventions: Device: Er:YAG Laser
- Carbon Fiber Curette (Active Comparator): Carbon fiber curette only
  Interventions: Other: Carbon Fiber Curette
- Er:YAG Laser + Carbon Fiber Curette (Experimental): Combination of Er:YAG Laser and carbon fiber curette
  Interventions: Device: Er:YAG Laser; Other: Carbon Fiber Curette
- No Treatment (No Intervention): No treatment (control)

INTERVENTIONS:
Device: Er:YAG Laser — Titanium disks will be decontaminated ex-vivo with the Er:YAG laser.
  Arms: Er:YAG Laser; Er:YAG Laser + Carbon Fiber Curette
Other: Carbon Fiber Curette — Titanium disks will be decontaminated ex-vivo with carbon fiber curettes
  Arms: Carbon Fiber Curette; Er:YAG Laser + Carbon Fiber Curette

SUMMARY:
The American Association of Oral and Maxillofacial Surgeons estimated that 69% of adults ages 35 to 44 have lost at least one permanent tooth. Dental implants have revolutionized dentistry by providing tooth-like replacement for missing teeth and a solution that is predictable with long-term success..

After the implant is placed, natural bacteria from the mouth can develop around implants just like around natural teeth. Studies have shown that bacterial contamination can cause peri-implantitis- gum disease or inflammation around the implant, eventually leading to bone loss. Removing bacteria from dental implant surfaces can prevent peri-implantitis, and surface debridement constitutes the basis of treatment of peri-implant disease.

Typically, mechanical hand instrumentation using curettes to remove biofilm and calculus is the main basis for periodontal therapy. However, total debridement is difficult, and the hand tools may damage the surface of the implant and making it more plaque retentive. Studies have shown that mechanical non-surgical therapy alone is not sufficient to treat peri-implantitis.

There is evidence that a dental laser may be an effective method to remove bacteria from implant surfaces, with less damage to the surface. One type of dental laser, Er:YAG, appears optimal for implant decontamination as the Er:YAG laser energy is primarily absorbed by water, resulting in vaporization of bacteria and minimal surface alterations on the implant surface.The aim of this study is to evaluate the efficiency of biofilm decontamination of Er:YAG laser compared to carbon fiber curette.

DETAILED DESCRIPTION:
The aim of this study is to compare the amount of residual biofilm on titanium discs after decontamination with Er:YAG laser and carbon fiber curette.

In the first phase of the study, custom mouth guards that holds multiple titanium discs will be fabricated. Experimental subjects will be instructed to wear this mouth guard for 72 hours, during which time a natural bacterial biofilm will form on the disc surfaces.

The second phase of the study will be performed ex vivo after collecting the discs from the subjects. Discs retrieved from each mouth guard will be randomized over the 4 treatment groups, so that each subject will contribute two discs to each treatment group: 1) Er:YAG laser, 2) carbon fiber curette, 3) combination of carbon fiber curette and Er:YAG laser, and 4) no treatment (control). The biofilm will be stained and the residual biofilm will be visualized under fluorescence microscopy. Statistical methods will be used to determine the significance of each treatment modality.

The primary outcome of the study is the percent area of the titanium disc covered by biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Presence of enough teeth to support the mouth guard.
* Subjects diagnosed with clinical health, gingivitis, or slight chronic periodontitis defined as periodontal inflammation with slight (1-2mm) attachment loss.

Exclusion Criteria:

* Subjects with insufficient dental support for the mouth guard
* Subjects diagnosed with moderate or severe chronic periodontitis.
* Subjects with known allergy to acrylic or titanium.
* Subjects who smoke cigarettes, cigars, snuff tobacco, or any other form of smoking.
* Subjects with a history of antibiotic treatment within the last six months.
* Subjects with contraindications to wearing a mouth guard, such as chronic obstructive pulmonary disease or severe sleep apnea.
* Subjects with uncontrolled or debilitating medical conditions, including but not limited to subjects with uncontrolled diabetes, hematologic disorders, cancers, immunosuppression, severe cardiovascular disease, or uncontrolled thyroid disease
* Subjects that are currently pregnant according to self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gyurko, DMD, PhD, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2017 to August 2018, 8 enrollments were made in the Department of Periodontology at Tufts University School of Dental Medicine
Pre-assignment Details: Each subject participates in each arm, as 2 titanium discs from each subject are distributed among all 4 arms.
Units Other Than Participants: 2 titanium disks per enrollee per arm
Groups:
- All Study Participants: Each participant provides 2 Titanium disks that are decontaminated ex-vivo with the Er:YAG laser, with carbon fiber curette, with titanium brush, or not decontaminated.
Period: Overall Study
Arm/Group | All Study Participants
Started | 8; 64 2 titanium disks per enrollee per arm
YAG Laser | 8; 16 2 titanium disks per enrollee per arm
Carbon Fiber Curette | 8; 16 2 titanium disks per enrollee per arm
Titanium Brush | 8; 16 2 titanium disks per enrollee per arm
Not Decontaminated | 8; 16 2 titanium disks per enrollee per arm
Completed | 8; 59 2 titanium disks per enrollee per arm
Not Completed | 0; 5 2 titanium disks per enrollee per arm

BASELINE CHARACTERISTICS:
Population: Each participant contributes 2 titanium discs to each arm therefore creating 64 discs to analyze across 4 arms.
Groups:
- All Study Participants: Titanium disks are decontaminated ex-vivo with the Er:YAG laser, with carbon fiber curettes, with titanium brush, or are not decontaminated .
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Indian | 1
  White | 1
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Bacteria Biofilm
Description: Percent area of the titanium disc covered by bacteria biofilm
Time Frame: 3 days
Population: From 64 collected titanium disks, 5 were removed from analysis. 4 disks were dislodged from 2 enrolled participants and 1 disk was excluded due to improper magnification of the SYTO 9 imaging.
Measure: Mean (Standard Deviation); unit: percentage of disc covered
Units Other Than Participants: Titanium disks
Groups:
- Laser: Titanium disks are decontaminated ex-vivo with the Er:YAG laser.
- Curette: Titanium disks are decontaminated ex-vivo with carbon fiber curettes
- Brush: Titanium disks are decontaminated ex-vivo with titanium brush
- Control: Titanium disks are not decontaminated
Arm/Group | Laser | Curette | Brush | Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
Number analyzed (Titanium disks) | 15 | 15 | 15 | 14
percentage of disc covered | 32.78 (24) | 20.14 (19.15) | 11.8 (10.29) | 74.03 (21.61)

ADVERSE EVENTS:
Time Frame: 3 days (the duration of wearing the intraoral appliance)
Arm/Group | Er:YAG Laser | Carbon Fiber Curette | Er:YAG Laser + Carbon Fiber Curette | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8 | 2/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Er:YAG Laser (N=8) | Carbon Fiber Curette (N=8) | Er:YAG Laser + Carbon Fiber Curette (N=8) | No Treatment (N=8)
Titanium disc dislodged from appliance (Product Issues) | 2 (2) | 2 (2) | 2 (2) | 2 (2) — Titanium discs were dislodged from the appliance in 2 of the 8 participants. Dislodged discs were excluded from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03100435/Prot_SAP_001.pdf